CLINICAL TRIAL: NCT02920372
Title: Generation of Positive Biological Samples to Epoetin for Doping Control.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Rafael de la Torre, PhD, Parc de Salut Mar
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IMIMFTCL/EPO; 2016-002866-29 (EudraCT Number)
Record Dates: First submitted 2016-09-29; First posted 2016-09-30 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: There Are no Conditions Under Study. Healthy Volunteers
MeSH Terms: interventions — Epoetin Alfa

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EPOETIN ALFA (Experimental)
  Interventions: Drug: EPOETIN ALFA

INTERVENTIONS:
Drug: EPOETIN ALFA

SUMMARY:
The study consists of generation of biological samples (in blood and urine) positive to Epoetin alfa for laboratories that wish to perform the analysis of doping controls and maintain accreditation from World Anti-Doping Agency.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male volunteers aged from 18 to 50 years.
2. A health profile devoid of organic or physiological disorders.
3. The ECG and general blood and urine laboratory tests performed before the study should be within normal ranges. Minor or occasional changes from normal ranges are accepted if, in the investigator's opinion, considering the current state of the art, they are not clinically significant, are not life-threatening for the subjects and do not interfere with the product assessment. These changes and their non-relevance will be justified in writing specifically.
4. Body mass index (BMI=weigh/height2) will range between 19 and 27 Kg/m2 and weight between 50 and 110 kg.
5. Understanding and accepting the study procedures and signing the informed consent form.

Exclusion Criteria:

1. Non compliance of the inclusion criteria.
2. Having suffered any organic disease or major surgery in the three months prior to start this study.
3. A prior history of or presence of significant cardiovascular, neurological, haematological, psychiatric, hepatic, gastrointestinal, pulmonary, endocrine, immunologic or renal disease that, in the investigator's opinion, considering the current state of the art, they are clinically significant, are life-threatening for the subjects and could interfere with the product assessment; or which may lead to suspecting a disorder in drug absorption, distribution, metabolism or excretion, or that suggest gastrointestinal irritation due to drugs.
4. History or clinical evidence of psychiatric disorders, alcoholism, drug abuse, or regular use of psychoactive drugs.
5. History of hypertension, seizures, endocrine disorders (such as diabetes and hypothyroidism), coagulation disorders, kidney and/or liver disease.
6. Subjects for which the drug involved in the study is counter indicated.
7. Smokers of more than 20 cigarettes per day.
8. Taking more than 35 g of alcohol per day.
9. Drinking more than 5 drinks containing xanthines per day.
10. Regular use of any drug in the month prior to the study sessions. The treatment with single or limited doses of symptomatic medicinal products in the week prior to the study sessions will not be a reason for exclusion if it is calculated that it has been cleared completely the day of the experimental session.
11. Have taken part in studies with blood donation in the last 8 weeks prior to start this study.
12. History of allergy, idiosyncrasy, hypersensitivity or adverse reactions to the active substance or any excipients.
13. Have been volunteer in another study with drugs in the last 3 months prior to start this study.
14. Subjects with positive serology for hepatitis B, C or HIV.
15. Subjects unable to understand the nature, consequences of the study and the procedures requested to be followed.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2016-11-30 (Actual); Primary Completion 2017-01-17 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Blood and urine concentrations of Epoetin alfa | From 48-72 hours pre-administration to 144 hours post administration
  Urine samples will be collected in different time periods: -48 to -24h, - 24h to 0h (pre-administration), 0 to 24h, 24 to 48h, 48 to 72h, 72 to 96h, 96 to 120h and 120 to 144h (post-administration). 10 mL of blood and dried blood spot (DBS) microvolume sampling with FTA DMPK -C cards will be collected at different time points: 48-72 hours before the first administration of the drug, before administration (0h, baseline), at 24, 48, 72 and 96 hours after administration of the drug. In session 5, blood samples will be collected at 0h (pre-administration) and at 1h, 4h and 8h after the administration of the drug.